CLINICAL TRIAL: NCT03679832
Title: Assessing the Impact of A Nutrition-Focused Quality Improvement Program in Hospitalized Malnourished Patients in an Academic University Hospital in Vietnam
Brief Title: A Nutrition-Focused Quality Improvement Program in Hospitalized Malnourished Patients
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Collaborators: University Medical Center, Vietnam (Unknown)
Responsible Party: Sponsor
Other Study IDs: HA32
Record Dates: First submitted 2018-08-17; First posted 2018-09-20 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Historical Group 1: Patients admitted at UMC between September 2015 and October 2016
- Historical Group 2: Patients admitted at UMC between November 2016 and up to the beginning of the QIP
- Nutrition-Focused QIP: Patients admitted at UMC that meet eligibility criteria and prospectively enrolled into QIP including malnutrition screening, nutrition consultation, expedited provision of oral nutritional supplementation (ONS) and encouragement of ONS consumption 30-days post discharge

SUMMARY:
This study includes pre and post-Quality Improvement Program groups. A nutrition-focused Quality Improvement Program will be implemented to assess the health and economic outcomes in malnourished hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at risk / malnourished, defined by an MST score ≥ 2 the first 24 hours post hospital admission
* Patients are admitted for the following diagnoses: Respiratory, Digestive Surgery, Cardiology, General Internal Medicine (including Endocrinology), and Gastrointestinal
* Patient is able to consume foods and beverages orally
* Patients with life expectancy ≥ 30 days
* Patient is literate and willing to voluntarily sign and date Informed Consent Form (ICF)

Exclusion Criteria:

* Subject has severe dementia or delirium and has no dedicated caregiver who could assure their compliance with QIP study requirements
* Subject has an eating disorder, history of significant neurological or psychiatric disorder, or other conditions that may interfere with study product consumption or compliance with study protocol procedures
* Subject is known to be allergic or intolerant to any ingredient found in the study products
* Subject is pregnant
* Subject is intubated, receiving tube feeding or parenteral nutrition

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a single-site in Vietnam meeting eligibility criteria for retrospective or prospective participation.
Sampling Method: Non-Probability Sample
Enrollment: 1670 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Hospital Length of Stay | From Date of Admission until Date of Discharge or Death from any cause, assessed through follow up (30-day Post Discharge)
  Chart Review

SECONDARY OUTCOMES:
Healthcare Resource Utilization | Hospital Admission to 30-day Post Discharge
  Chart Review

CONTACTS AND LOCATIONS:
Overall Officials: Suela Sulo, PhD,MSc, Study Chair — Abbott Nutrition
Locations (1):
- University Medical Center, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided